CLINICAL TRIAL: NCT05348668
Title: Hybrid Dose-fraction Radiotherapy for Metastatic Driven-genes Negative Non-small Cell Lung Cancer: A Phase II Multi-institutional Study
Brief Title: Hybrid Dose-fraction Radiotherapy for Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Dong Qian, Professor, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-ky301
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: metastatic driven-genes negative non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: 74 patients with metastatic driven-genes negative non-small cell lung cancer to receive the combination of hybrid dose-fraction radiotherapy with ICI
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hybrid dose-fraction Radiotherapy Arm (Experimental): Patients in this arm would receive hybrid dose-fraction radiotherapy combined with immune checkpoint inhibitors.
  Interventions: Drug: Hybrid dose-fraction Radiotherapy combined with immune checkpoint inhibitors

INTERVENTIONS:
Drug: Hybrid dose-fraction Radiotherapy combined with immune checkpoint inhibitors — Hybrid dose-fraction Radiotherapy combined with immune checkpoint inhibitors
  Other Names: no other interventions

SUMMARY:
The combination of immune checkpoint inhibitors (ICI) and local ablative radiotherapy has been demonstrated to be able to increase the survival of patients with metastatic driven-genes negative non-small cell lung cancer. Various dose-fraction of radiotherapy could exert different effects on the immune system. Ablative-dose could induce immunogenic cell death through the activation of CD8+(Cluster of Differentiation) T cells. Low-dose could modulate immune microenvironment from immunosuppression to inflammatory anti-tumor phenotype. This trial is designed to validation the safety and primary efficacy of the combination of hybrid dose-fraction radiotherapy with ICI for metastatic driven-genes negative non-small cell lung cancer patients.

DETAILED DESCRIPTION:
Trial Title: Hybrid dose-fraction Radiotherapy for metastatic driven-genes negative non-small cell lung cancer: A phase II multi-institutional study Trial Objective: To explore the safety and primary efficacy of the combination of hybrid dose-fraction radiotherapy with ICI for metastatic driven-genes negative non-small cell lung cancer patients.

Trial Design: This trial is designed to enroll 74 patients with metastatic driven-genes negative non-small cell lung cancer to receive the combination of hybrid dose-fraction radiotherapy with ICI.

Staging Examination before Radiotherapy: a. ECOG scoring. b. Cranial contrast MRI and PET-CT (Positron Emissions Tomography), or cranial contrast MRI (preferred), chest contrast CT, abdominal ultrasonography and bone scan. c. Bronchoscopy for centrally located lung cancer.

Inductive therapy ICI±chemotherapy for 4-6 cycles. Pembrolizumab and Tislelizumab are preferred. Chemotherapy regimens could be referred to NCCN (National Comprehensive Cancer Network) guidelines.

Restaging examination after inductive therapy is mandatory: a. ECOG scoring. b. Cranial contrast MRI, chest contrast CT, abdominal ultrasonography.

Patients with disease PR or SD (RECIST v1.1) evaluated by restaging after inductive therapy could be included into this trial. Patients would receive hybrid dose-fraction radiotherapy and ICI maintenance.

Radiotherapy CT Simulation: CT with intravenous contrast is recommended for simulation. Scan thickness should be less than 5 mm from lower margin of mandibular to lower margin of L2. For pulmonary lesions, 4D-CT (Four-Dimensional CT) localization is recommended.

Delineation of Targets:

For patients with oligometastasis, including synchronous oligometastatic disease & metachronous oligorecurrence, all lesions should be prescribed with an ablative dose. The dose-fraction modalities are as following:

Thoracic lesions: 50Gy/5f (50 Gray/5 fractions), 60Gy/8f, 60Gy/15f, 48Gy/12f. Intracranial lesions: 30Gy/10f (Whole Brain Irradiation), 30Gy/3f, 30Gy/5f, 45Gy/15f.

Hepatic lesions: 50Gy/5f, 40Gy/5f, 32Gy/4f. Adrenal lesions: 50Gy/5f, 40Gy/5f, 32Gy/4f. Osseous lesions: 27Gy/3f, 40Gy/5f, 30Gy/5f, 39Gy/13f. Other lesions: Refer to the above dose-fraction. For patients with systemic metastasis, high-dose should be prescribed to 1-3 lesions (longest diameter>1cm). All of the remaining lesions should be given low-dose. High-dose includes 24-40Gy/3-5f. Low-dose includes 6-15Gy/4-10f.

The Planning Target Volume (PTV) was defined as an 8-mm margin of the GTV (Gross Tumor Volumn) for tumor motion and set-up variations.

The delivery of ablative dose and high-dose should utilize the technology of SABR (Stereotactic Ablative Body Radiotherapy).

Dosimetric Limitation of Organ at Risk: 95% prescription dose should cover 100% PTV and 95% PTV should receive 100% prescription dose.

The dose constraints of organs at risk could refer to TG 101 (Task Group 101) report.

Treatment Implementation: Radiotherapy is implemented every day. Cone-beam CT should be utilized every day to minimize set-up error.

Follow-up: Patients should be follow-up every three months right after the completion of radiotherapy to disease progression.

Primary Endpoint: Progress-free Survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old;
* Eastern Cooperative Oncology Group (ECOG) 0-1;
* Non-small cell lung cancer, including squamous-cell carcinoma, adenocarcinoma, large-cell carcinoma, adenosquamous carcinoma;
* Stage IVA and IVB confirmed by radiological examination (AJCC 8th Edition);
* Driven-genes negative including EGFR (Epidermal Growth Factor Receptor), ALK (Anaplastic Lymphoma Kinase), ROS1 (ROS Proto-Oncogene 1), KRAS G12C (Kirsten Rat Sarcoma Viral Oncogene), BRAF V600E (v-raf murine sarcoma viral oncogene homolog B1), MET exon14 (Mesenchymal Epithelial Transition Factor), RET (Rearranged during Transfection Proto-oncogene), NTRK1/2/3 (NeuroTrophin Receptor Kinase);
* First-line treatment of ICI±chemotherapy;
* Partial response (PR) or stable (SD) after first-line treatment;
* Signature of inform consent.

Exclusion Criteria:

* younger than 18 years old or older than 75 years old;
* ECOG>1;
* Small-cell lung cancer and other neuroendocrine carcinoma;
* Non stage IV confirmed by radiological examination;
* Driven-genes positive including EGFR, ALK, ROS1, KRAS G12C, BRAF V600E, MET exon14, RET, NTRK1/2/3;
* First-line treatment of other therapy rather than ICI±chemotherapy;
* Complete response (CR) or progression (PD) after first-line treatment;
* Contraindications for radiotherapy, chemotherapy and ICI;
* No signature of inform consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival | 1-year
  Progression-free Survival evaluated by RECIST (v1.1)

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provicial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No